CLINICAL TRIAL: NCT06730568
Title: Effect of Different Non-surgical Treatment Approaches of Peri-implantitis: a Multi-arm Randomized Controlled Clinical Trial
Brief Title: Effect of Different Non-surgical Treatment Approaches of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Nihal ERAYDIN, Assistant Professor, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-RCT
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Peri-implant Inflammation; Peri-Implantitis and Peri-implant Mucositis; Non-surgical Treatment
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Mechanical Instrumentation (M) (Active Comparator): The participants in the mechanical instrumentation (M) group were treated with conventional submarginal instrumentation using titanium curettes.
  Interventions: Procedure: Submarginal mechanical instrumentation
- Mechanical Instrumentation with Chlorhexidine (MC) (Experimental): Participants in the mechanical instrumentation with chlorhexidine (MC) group were treated with conventional submarginal instrumentation using titanium curettes followed by adjunctive chlorhexidine irrigation.
  Interventions: Procedure: Submarginal mechanical instrumentation and chlorhexidine irrigation
- Mechanical Instrumentation with Ozone (MO) (Experimental): Participants in the mechanical instrumentation with chlorhexidine (MC) group were treated with conventional submarginal instrumentation using titanium curettes followed by gaseous ozone
  Interventions: Procedure: Submarginal mechanical instrumentation and ozone application
- Mechanical Instrumentation with Air Abrasion (MA) (Experimental): The participants in the mechanical instrumentation with glycine powder air abrasion (MA) group were treated with conventional submarginal instrumentation using titanium curettes and followed by adjunctive glycine air-abrasion.
  Interventions: Procedure: Submarginal mechanical instrumentation and air abrasion
- Air Abrasion Monotherapy (A) (Experimental): The participants in the air abrasion monotherapy (A) group were treated exclusively with glycine powder-based air abrasion.
  Interventions: Procedure: Air abrasion monotherapy

INTERVENTIONS:
Procedure: Submarginal mechanical instrumentation — Local anesthesia was applied before the procedure. The operator performed submarginal mechanical debridement until the implant surface was deemed adequately cleaned. No adjunctive therapies were applied in this group.
  Arms: Mechanical Instrumentation (M)
Procedure: Submarginal mechanical instrumentation and chlorhexidine irrigation — The participants in the mechanical instrumentation with chlorhexidine (MC) group were treated with conventional submarginal instrumentation using titanium curettes. Local anesthesia was applied before the procedure. The operator performed submarginal mechanical debridement until the implant surface was deemed adequately cleaned. Following mechanical instrumentation, the peri-implant pockets were irrigated with 0.2% chlorhexidine digluconate solution for 1 minute.
  Arms: Mechanical Instrumentation with Chlorhexidine (MC)
Procedure: Submarginal mechanical instrumentation and ozone application — The participants in the mechanical instrumentation with ozone (MO) group were treated with conventional submarginal instrumentation using titanium curettes. Local anesthesia was applied before the procedure. The operator performed submarginal mechanical debridement until the implant surface was deemed adequately cleaned. Following mechanical instrumentation, gaseous ozone was applied to the peri-implant pockets using an ozone-generating device and a specialized glass fiber probe. The ozone gas was delivered to four sites (mesial, distal, buccal, and lingual) for 15 seconds per site, resulting in a total application time of 1 minute per implant. The device operated at a power of 3 watts and 80% oxygen concentration, as recommended by the manufacturer.
  Arms: Mechanical Instrumentation with Ozone (MO)
Procedure: Submarginal mechanical instrumentation and air abrasion — The participants in the mechanical instrumentation with glycine powder air abrasion (MA) group were treated with conventional submarginal instrumentation using titanium curettes. Local anesthesia was applied before the procedure. The operator performed submarginal mechanical debridement until the implant surface was deemed adequately cleaned. Following mechanical instrumentation, the peri-implant pockets were treated with glycine powder-based air abrasion using an air-abrasion device (AIR-FLOW® handy 3.0 PERIO HANDPIECE, EMS, Nyon, Switzerland) and a flexible Perio-Flow® nozzle. The nozzle was inserted into the pockets and guided in a circular motion from coronal to apical, parallel to the implant surface, in a non-contact mode as recommended by the manufacturer. The air-abrasion treatment was applied to four sites (mesial, distal, buccal, and lingual) for 5 seconds per site, resulting in a total application time of 20 seconds per implant.
  Arms: Mechanical Instrumentation with Air Abrasion (MA)
Procedure: Air abrasion monotherapy — The participants in the glycine powder air abrasion monotherapy (A) group were treated exclusively with glycine powder-based air abrasion. Local anesthesia was applied before the procedure. The peri-implant pockets were instrumented with an air-abrasion device using glycine powder and a flexible nozzle. The nozzle was inserted into the pockets and guided in a circular motion from coronal to apical, parallel to the implant surface, in a non-contact mode as recommended by the manufacturer. The air-abrasion treatment was applied to four sites (mesial, distal, buccal, and lingual) for 5 seconds per site, resulting in a total application time of 20 seconds per implant. .
  Arms: Air Abrasion Monotherapy (A)

SUMMARY:
Peri-implantitis is a biofilm-associated pathological condition characterized by inflammation within the peri-implant mucosa, which leads to the progressive loss of the surrounding supporting bone tissue. The primary goal of managing peri-implantitis is to control the peri-implant biofilm and resolve inflammation. Nonsurgical treatment of peri-implantitis by submarginal mechanical instrumentation alone typically provides clinical improvements, particularly in non-advanced cases. However, to ensure surface decontamination and enhance treatment outcomes, alternative or adjunctive methods, such as systemic/local antibiotics, antiseptics, lasers, and air-abrasion systems, have been proposed.

Therefore, the null hypothesis (H0) of the present study is that no statistically significant difference would be detected in clinical inflammation signs among patients diagnosed with early-stage peri-implantitis after undergoing one of the following treatments: nonsurgical mechanical instrumentation alone, mechanical instrumentation plus chlorhexidine (CHX), mechanical instrumentation plus gaseous ozone, mechanical instrumentation plus glycine air polishing, or glycine air polishing alone.

ELIGIBILITY:
Inclusion Criteria:

* the presence of at least one titanium implant with clinical and radiographic signs of initial to moderate peri-implantitis
* single-unit or partial restorations without overhangings
* absence of occlusal overload
* the presence of at least 2 mm of keratinized attached peri-implant mucosa
* periodontally healthy participants with a good level of oral hygiene

Exclusion Criteria:

* the presence of implant mobility
* systemic diseases (i.e. diabetes (HbA1c <7), osteoporosis, bisphosphonate medication) which could affect the outcome of treatment
* smoking
* placement, and prosthetic loading of implants within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Probable Pocket Depth | Baseline, 3 months, and 6 months after treatment

SECONDARY OUTCOMES:
Bleeding on Probing | Baseline, 3 months, and 6 months after treatment
Plaque Index | Baseline, 3 months, and 6 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Dentistry Faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No